CLINICAL TRIAL: NCT00058214
Title: A Phase II Trial of Perifosine (IND 58,156; NSC# 639966) in Biochemically Recurrent, Hormone Sensitive Prostate Cancer
Brief Title: Perifosine in Treating Patients With Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet interim stopping criteria for continuation to the second stage.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02832; PHII-44; N01CM17101 (NIH); CDR0000287195 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perifosine; octadecyl-(N,N-dimethylpiperidino-4-yl)-phosphate

ARMS (1):
- Treatment (perifosine) (Experimental): Patients receive oral perifosine once daily on days 1-28. On day 1 of course 1 only, patients receive 2 doses of oral perifosine. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease by PSA alone may receive up to 3 additional courses of therapy after documentation of progression.
  Interventions: Drug: perifosine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: perifosine — Given orally
  Other Names: D21266; octadecylphosphopiperidine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of perifosine in treating patients who have recurrent prostate cancer. Drugs used in chemotherapy such as perifosine use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the PSA response in prostate cancer patients with only biochemical recurrence after local curative therapy who are then treated with perifosine.

II. To assess the secondary endpoints of a) six-month increase in PSA levels compared to baseline, b) PSA doubling time and c) time to PSA progression in prostate cancer patients receiving perifosine.

III. To evaluate the qualitative and quantitative toxicities of this agent in this patient population.

IV. To investigate potential molecular markers predictive of decreased PSADT and possibly PSA response in prostate cancer patients receiving perifosine.

OUTLINE: This is a multicenter study. Patients are stratified according to prior therapy (surgery vs radiotherapy with or without brachytherapy vs surgery and radiotherapy) and original combined Gleason score (7 or less vs 8-10).

Patients receive oral perifosine once daily on days 1-28. On day 1 of course 1 only, patients receive 2 doses of oral perifosine. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease by PSA alone may receive up to 3 additional courses of therapy after documentation of progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Patients must have a rising PSA >= 2.0 following a nadir after local curative therapy (either radical prostatectomy and/or pelvic radiation) with no clinical or radiographic evidence of metastatic disease; PSA >= 2.0 elevation must be confirmed by two consecutive increases, each measured at least 2 weeks apart; only patients with a biochemical (PSA) recurrence with no physical exam or radiographic evidence of local or distant relapse are eligible
* Prior hormonal therapy in the form of neoadjuvant or adjuvant therapy is allowed as long as neither lasted for more than 9 months; androgen deprivation therapy must have been completed at least one year prior to registration; patients could not have had a rising PSA at the time that neoadjuvant or adjuvant therapy was stopped
* Life expectancy of greater than 3 months
* Karnofsky performance status > 60%
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,00/uL
* Total bilirubin =< 1.5 mg/dL
* AST (SGOT)/ALT (SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min
* Computed tomography scan or MRI of the pelvis negative for metastatic disease within 3 months prior to registration
* Bone scan negative for metastatic disease within 3 months prior to registration
* Chest PA and lateral films negative for metastatic disease within 3 months prior to registration
* Prior vaccine therapy is allowed if completed at least 6 months prior to registration
* Men enrolled in this trial must agree to use adequate contraception prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had any prior cytotoxic chemotherapy
* Patients may not be receiving any other investigational agents
* Patients receiving concurrent chemotherapeutic agents, biological response modifiers, radiation therapy, corticosteroid or hormonal therapy; no complementary or alternative therapy (e.g., St. John's Wort, PC-SPES, or any other herbal remedies taken for the purpose of treating prostate cancer) may be given during protocol treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine
* Androgen deprivation given for reasons other than neoadjuvant or adjuvant therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of any site, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Perifosine): Patients receive oral perifosine 100 mg once daily on days 1-28. On day 1 of course 1 only, patients receive 2 doses of oral perifosine at 450 mg. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease by PSA alone may receive up to 3 additional courses of therapy after documentation of progression.
  perifosine: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Perifosine)
Started | 25
Completed | 24
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Perifosine)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 67 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: A PSA normalization (PSA-N) - was recorded on case report forms for any evaluation in which the PSA level was undetectable (< 0.1 ng/mL). If the PSA-N response was confirmed by a second measurement ≥ 4 weeks later, the patient's best PSA response was considered PSA-N. PSA-PR was recorded if the PSA decreased by ≥ 50% from baseline (pretreatment) values and confirmed by a second measurement ≥ 4 weeks later. PSA-PD was recorded upon the appearance of ≥ 1 new lesion on radiographs consistent with metastatic disease, an absolute increase in PSA value of 5 ng/mL relative to the lowest postenrollment PSA value (including the baseline PSA value), or if the PSA doubling time was < 2 months. PSA-SD constituted responses that did not qualify for PSA-N, PSA-PR, or PSA-PD. Response = PSA-N + PSA-PR.
Time Frame: Up to 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Perifosine)
Number analyzed (Participants) | 24
percentage of participants | 0

2. Secondary Outcome: Time to Progression
Description: Estimated using the product-limit method of Kaplan and Meier. Progression was defined as the appearance of ≥ 1 new lesion on radiographs consistent with metastatic disease, an absolute increase in PSA value of 5 ng/mL relative to the lowest postenrollment PSA value (including the baseline PSA value), or if the PSA doubling time was < 2 months.
Time Frame: From the date of registration to the date of documented PSA progression, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Perifosine)
Number analyzed (Participants) | 25
months | 6.64 [4.53 to 12.81]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 60 month period.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Perifosine)
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Perifosine) (N=25)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Perifosine) (N=25)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (20)
Palpitations (Cardiac disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 16 (27)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 3 (8)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (13)
(Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chest pain (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 12 (17)
General symptom (General disorders) | 2 (2)
Oedema NOS (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Infection, Viral (COH) (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (7)
Creatinine increased (Investigations) | 2 (2)
Hyperbilirubinemia (Investigations) | 1 (2)
Hypercholesterolemia (Investigations) | 1 (2)
Leukopenia (Investigations) | 2 (9)
Lymphopenia (Investigations) | 4 (8)
Neutrophil count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (28)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (7)
Headache (Nervous system disorders) | 2 (4)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (10)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less